CLINICAL TRIAL: NCT01488565
Title: A Single Arm Pilot Study of Azacitidine in Myelodysplastic Syndrome / Acute Myeloid Leukaemia, With Eltrombopag Support for Thrombocytopenia.
Brief Title: A Single Arm Pilot Study of Azacitidine in Myelodysplastic Syndromes (MDS) / Acute Myeloid Leukaemia (AML), With Eltrombopag Support for Thrombocytopenia
Acronym: Aza-E
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Collaborators: GlaxoSmithKline (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10/78
Record Dates: First submitted 2011-11-29; First posted 2011-12-08 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-02

CONDITIONS: Myelodysplastic Syndromes (MDS); Acute Myeloid Leukaemia (AML)
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Azacitidine; eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Azacitidine and Eltrombopag (Experimental): Vidaza (azacitidine) Revolade (eltrombopag)
  Interventions: Drug: Azacitidine and eltrombopag

INTERVENTIONS:
Drug: Azacitidine and eltrombopag — Standard: azacitidine D1-5, 8&9, until loss of clinical benefit. Experimental: eltrombopag at a dose ranging from 50-300mg for 6 months, continuing only in those deriving clinical benefit.
  Other Names: Vidaza (azacitidine); Revolade (eltrombopag)

SUMMARY:
Myelodysplastic Syndrome (MDS) is a disease of the bone marrow characterized by anemia,neutropenia, and thrombocytopenia (low red blood cell, white blood cell, and platelet counts). MDS patients with thrombocytopenia who fail standard therapies require regular platelet transfusions which are expensive and inconvenient, and are a risk for further serious bleeding complications. The new treatment of MDS using azacitidine has shown to increase the survival rate of MDS patients including to improve platelet production over time. However,in the early cycles of treatment with azacitidine,the low platelet counts tend to exacerbate before they provide any clinical benefit.

Eltrombopag is a drug designed to activate the thrombopoietin receptor. Eltrombopag has been able to increase platelet counts in healthy Thrombocytopenia Purpura (ITP), a disease where patients destroy their own platelets very rapidly and thus develop thrombocytopenia.

Eltrombopag is administered orally and is Therapeutic Goods Administration (TGA) approved for the treatment of thrombocytopenia in patients with chronic ITP who failed to respond to standard treatment.

This study is a single arm pilot study to evaluate the safety and tolerability of Eltrombopag in the treatment of low platelet counts in adult subjects with MDS treated using azacitidine This study also incorporates a correlative laboratory component designed to determined the mechanism of action of 5-azacitidine +/- Eltrombopag and to determine a baseline profile which may predict those most responsive. These studies will incorporate gene methylation and expression, and immunoprofiling.

ELIGIBILITY:
Inclusion Criteria:

* Patients with low platelet count (<=150 x109/L)and in addition disease diagnosis of either MDS, or nonproliferative CMML or low marrow blast count AML not suitable for induction chemotherapy
* Age >18 years
* ECOG score 0-2 at screening
* Life expectancy ≥12 weeks
* Ability to comply with the adequate contraception in patients of childbearing potential.

Exclusion Criteria:

* Subjects with the diagnosis acute promyelocytic leukaemia
* Prior treatment with azacitidine or any other methyl-transferase inhibitor (e.g. decitabine)
* Prior treatment with eltrombopag, romiplostim, or other TPO-receptor agonist
* AML or MDS requiring cytoreductive therapy (eg hydroxyurea, ara-c, thioguanine etc) in the month prior to study entry
* Known uncontrolled medical conditions which may compromise participation in this study including but not limited to:

  * Poorly controlled congestive heart failure: ejection fraction <30% measured in past 6 months) or NYHA class IV
  * Arrhythmia known to increase the risk of thromboembolic events.
  * Unstable angina or an ischaemic cardiac event requiring hospital admission in the previous 12 months.
  * Unresolved GI disease that may significantly alter the absorption of eltrombopag
* Known pro-thrombotic condition as defined by a history ≥1 unprovoked deep venous thrombosis or pulmonary embolism, or any DVT/PE with a procoagulant condition screen suggesting the presence of a procoagulant condition (prothrombin gene mutation homozygosity, factor V leiden homozygosity, antithrombin deficiency, lupus anticoagulant syndrome).
* History of Ischaemic neurological event (TIA or stroke) within the preceding 2 years.
* Inadequate renal function (eGFR <30 ml/min by Cockcroft-Gault (C-G) formula, or as measured by 24 hour urinary creatinine clearance)
* Inadequate hepatic function:

  * bilirubin ≥1.5xULN - ≤80µmol/L acceptable if attributed to haemolysis, ineffective erythropoiesis or iron overload). This applies also for patients with Gilbert's Syndrome.
  * AST or ALT ≥2xULN (≤3xULN acceptable if attributed to transfusion-associated iron overload)
  * Patients with known liver cirrhosis.
* Other concurrent severe and/or uncontrolled medical conditions including a history of malignancy other than MDS/AML in the preceding 2 years requiring chemotherapy and/or radiotherapy. Non melanotic skin cancers requiring low dose local radiotherapy or topical agents are allowed on study if considered clinically stable or healed.
* Women who are pregnant or breast-feeding.
* Treatment with growth factors such as erythropoietin, GCSF or stem cell factor in the 21 days prior to commencement of study therapy.
* Active or uncontrolled infections.
* Subjects with known HIV infection.
* Has any other clinically important abnormalities as determined by the investigator that may interfere with his or her participation in or compliance with the study
* Bone marrow fibrosis that leads to an inability to aspirate marrow for quality cytological assessment, termed a "dry tap".
* Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule. This condition must be discussed with the patient prior to signing consent and registration in the trial.
* Splenomegaly >14cm on the screening ultrasound examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-12; Primary Completion 2014-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Number of events of non-haematological toxicities related to the combination of eltrombopag and azacitidine | At 6 cycles of therapy (approx 6 months)
  The number of events of Grade III/IV non-haematological toxicities will be measured based on the possibly, probably or definitely relatedness to the combination of eltrombopag and azacitidine

SECONDARY OUTCOMES:
Number of patients with improved platelet counts and the dose at which this may be achieved. | Approximately 2.5 years after the last accrued patient completes study treatment
Correlation of the laboratory findings with the response of the combination of 5-azacitidine and eltrombopag in patients with MDS and low marrow blast count AML | Approximately 2.5 years after last accrued patient completes study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dickinson, Dr, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (2):
- Australia (2):
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - Cabrini Hospital, Malvern, Victoria